CLINICAL TRIAL: NCT02325531
Title: SPREAD-NET: PRactices Enabling Adapting and Disseminating in the Safety NET
Acronym: SPREAD-NET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); OCHIN, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01HL120894-01 (NIH); 1R01HL120894-01 (NIH)
Record Dates: First submitted 2014-12-15; First posted 2014-12-25 (Estimated); Results first posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus; Cardiovascular Disease
Keywords: implementation strategies; diabetes mellitus; cardiovascular disease; community health centers; quality improvement; translational medical research
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Clinics were randomized and data was collected at the clinic level, there was no data collected at the participant level.
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low support (Other): In this pragmatic comparative effectiveness trial, clinics NOT patients were randomized. Clinics were randomly assigned to one of the arms and support was provided to the clinic, not the patient.
  EHR-based toolkit Basic webinar
  Interventions: Other: Low support
- Medium support (Other): In this pragmatic comparative effectiveness trial, clinics NOT patients were randomized. Clinics were randomly assigned to one of the arms and support was provided to the clinic, not the patient.
  Support provided to the low support arm, PLUS Staff training Adaptive webinars
  Interventions: Other: Medium support
- High support (Other): In this pragmatic comparative effectiveness trial, clinics NOT patients were randomized. Clinics were randomly assigned to one of the arms and support was provided to the clinic, not the patient.
  Support provided to the low and medium support arms, PLUS Practice facilitation
  Interventions: Other: High support
- Comparison (Other): In this pragmatic comparative effectiveness trial, clinics NOT patients were randomized. Clinics were randomly assigned to one of the arms and support was provided to the clinic, not the patient.
  No support was provided by the researchers. The EHR-based toolkit was available to all clinics in the network if they actively searched it out in the EHR.
  Interventions: Other: Comparison

INTERVENTIONS:
Other: Low support — EHR-based tools, built by OCHIN, activated during Year 1 TOOLKIT, paper and electronic form, includes documents to help support ALL implementation, and
  BASIC WEBINAR, Annual, 1-hour, topics such as:
  Talking to Clinicians About ALL, Using The Monthly Feedback Report and Integrating the Toolkit into Workflows
  Arms: Low support
Other: Medium support — Same as provided to the low support arm, PLUS
  * STAFF TRAINING (2-day meeting in Portland, Oregon, Led by Implementation Specialists (IS), How to use the toolkit and how to train others to use it, Content guided by previous research, baseline survey results, study team and the S-N advisory group
  * ADAPTIVE WEBINARS, Quarterly 1-hr webinars, Content from basic webinars, tailored to topics requested by study clinics. Forum for group discussion and best practice sharing. Open any interested clinics in Arm 2 & 3.
  Arms: Medium support
Other: High support — Same as provided to the low and medium support arms, PLUS
  - PRACTICE FACILITATION: Site visits with support as needed, Staff presentations, Coaching on tools (how to present to clinic staff and how to use in the clinic workflow), Tailored problem-solving support to address identified barriers, Clinical questions fielded by RN practice facilitator and site clinician champion.
  Arms: High support
Other: Comparison — No support was provided by the researchers. The EHR-based toolkit was available to all clinics in the network if they actively searched it out in the EHR.
  Arms: Comparison

SUMMARY:
The investigators propose to compare the effectiveness of 3 strategies (low, medium, high intensity) at supporting CHCs' implementation of the ALL Initiative (an intervention shown to reduce patients' cardiovascular disease (CVD) event risk), through a cluster-randomized trial.

DETAILED DESCRIPTION:
The investigators propose to compare the effectiveness of 3 support strategies for optimizing the sustainable implementation of the evidence-based ALL intervention. To do so, the investigators will randomize 30 community health centers (CHCs) to receive 1 of 3 implementation support strategies: Low support (toolkit only), Medium (toolkit, staff training), High (toolkit, training, on-site facilitation). The study aims are as follows:

Aim 1: Compare the effectiveness of the 3 strategies (low, medium, high intensity) at supporting CHCs' implementation of the ALL intervention, through a cluster-randomized trial.

Hypothesis: Clinics randomized to receive more implementation support will be more likely than those randomized to receive less support (high>medium>low) to significantly improve the percent of their patients with (i) guideline-appropriate prescriptions for ACE/ARBs and statins, and (ii) last blood pressure (BP) and low-density lipoprotein (LDL) under control).

Aim 2: Assess how effectively the 3 strategies support intervention sustainability at 12, 24 and 36 months post-implementation, measured as maintenance of change over time (outcomes as in Aim 1).

Hypothesis: Clinics randomized to receive more implementation support will be more likely to maintain changes in the outcomes of interest.

Aim 3: Identify clinic characteristics associated with the support strategies' effectiveness (e.g. decision-making structures, leadership support, team processes / characteristics, readiness and capacity for change).

Research questions: What are the characteristics of clinics that achieve sustained change even with less implementation support, and of those that do not achieve change even with more support?

ELIGIBILITY:
Inclusion Criteria:

* Convenience sample, all patients with Diabetes Mellitus from 30 community health clinics (CHCs) that are members of OCHIN, Inc.

Exclusion Criteria:

* Patients without diagnosed DM

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Gold, PhD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente - Center for Health Research, Portland, Oregon, United States

REFERENCES:
- [Result] Gold R, Bunce A, Cowburn S, Davis JV, Nelson JC, Nelson CA, Hicks E, Cohen DJ, Horberg MA, Melgar G, Dearing JW, Seabrook J, Mossman N, Bulkley J. Does increased implementation support improve community clinics' guideline-concordant care? Results of a mixed methods, pragmatic comparative effectiveness trial. Implement Sci. 2019 Dec 5;14(1):100. doi: 10.1186/s13012-019-0948-5. PMID 31805968
- [Derived] Gruss I, Bunce A, Davis J, Gold R. Unintended consequences: a qualitative study exploring the impact of collecting implementation process data with phone interviews on implementation activities. Implement Sci Commun. 2020 Nov 4;1(1):101. doi: 10.1186/s43058-020-00093-7. PMID 33292848
- [Derived] Bunce AE, Gruss I, Davis JV, Cowburn S, Cohen D, Oakley J, Gold R. Lessons learned about the effective operationalization of champions as an implementation strategy: results from a qualitative process evaluation of a pragmatic trial. Implement Sci. 2020 Oct 1;15(1):87. doi: 10.1186/s13012-020-01048-1. PMID 32998750
- [Derived] Gold R, Hollombe C, Bunce A, Nelson C, Davis JV, Cowburn S, Perrin N, DeVoe J, Mossman N, Boles B, Horberg M, Dearing JW, Jaworski V, Cohen D, Smith D. Study protocol for "Study of Practices Enabling Implementation and Adaptation in the Safety Net (SPREAD-NET)": a pragmatic trial comparing implementation strategies. Implement Sci. 2015 Oct 16;10:144. doi: 10.1186/s13012-015-0333-y. PMID 26474759

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this pragmatic comparative effectiveness trial, clinics NOT patients were randomized. Clinics were randomly assigned to one of the arms and support was provided to the clinic, not the patient. No patients were recruited or consented.
Pre-assignment Details: Data was collected at the clinic level, there was no data collected at the participant level and therefore there are no participant numbers available for any results modules.
Units Other Than Participants: Clinics
Groups:
- Low Support: In this pragmatic comparative effectiveness trial, clinics NOT patients were randomized. Clinics were randomly assigned to one of the arms and support was provided to the clinic, not the patient.
  EHR-based toolkit Basic webinar
  Low support: EHR-based tools, built by OCHIN, activated during Year 1 TOOLKIT, paper and electronic form, includes documents to help support ALL implementation, and
  BASIC WEBINAR, Annual, 1-hour, topics such as:
  Talking to Clinicians About ALL, Using The Monthly Feedback Report and Integrating the Toolkit into Workflows
- Medium Support: In this pragmatic comparative effectiveness trial, clinics NOT patients were randomized. Clinics were randomly assigned to one of the arms and support was provided to the clinic, not the patient.
  Support provided to the low support arm, PLUS Staff training Adaptive webinars
  Medium support: Same as provided to the low support arm, PLUS
  * STAFF TRAINING (2-day meeting in Portland, Oregon, Led by Implementation Specialists (IS), How to use the toolkit and how to train others to use it, Content guided by previous research, baseline survey results, study team and the S-N advisory group
  * ADAPTIVE WEBINARS, Quarterly 1-hr webinars, Content from basic webinars, tailored to topics requested by study clinics. Forum for group discussion and best practice sharing. Open any interested clinics in Arm 2 & 3.
- High Support: In this pragmatic comparative effectiveness trial, clinics NOT patients were randomized. Clinics were randomly assigned to one of the arms and support was provided to the clinic, not the patient.
  Support provided to the low and medium support arms, PLUS Practice facilitation
  High support: Same as provided to the low and medium support arms, PLUS
  - PRACTICE FACILITATION: Site visits with support as needed, Staff presentations, Coaching on tools (how to present to clinic staff and how to use in the clinic workflow), Tailored problem-solving support to address identified barriers, Clinical questions fielded by RN practice facilitator and site clinician champion.
- Comparison: In this pragmatic comparative effectiveness trial, clinics NOT patients were randomized. Clinics were randomly assigned to one of the arms and support was provided to the clinic, not the patient.
  No support was provided by the researchers. The EHR-based toolkit was available to all clinics in the network if they actively searched it out in the EHR.
  Comparison: No support was provided by the researchers. The EHR-based toolkit was available to all clinics in the network if they actively searched it out in the EHR.
Period: Overall Study
Arm/Group | Low Support | Medium Support | High Support | Comparison
Started | NA; 9 Clinics (Data was collected at the clinic level, there was no data collected at the participant level) | NA; 11 Clinics (Data was collected at the clinic level, there was no data collected at the participant level) | NA; 9 Clinics (Data was collected at the clinic level, there was no data collected at the participant level) | NA; 137 Clinics (Data was collected at the clinic level, there was no data collected at the participant level)
Completed | NA; 9 Clinics (Data was collected at the clinic level, there was no data collected at the participant level) | NA; 11 Clinics (Data was collected at the clinic level, there was no data collected at the participant level) | NA; 7 Clinics (Data was collected at the clinic level, there was no data collected at the participant level) | NA; 137 Clinics (Data was collected at the clinic level, there was no data collected at the participant level)
Not Completed | NA; 0 Clinics | NA; 0 Clinics | NA; 2 Clinics | NA; 0 Clinics

BASELINE CHARACTERISTICS:
Population: This is a clinic randomized trial. No patients were recruited or consented in this study. Clinics were recruited and the intervention was conducted at the clinic level. Baseline data was collected on clinic rates. Only aggregate level data (percent of the population) was collected and it applied to clinics, not individuals.
Units Other Than Participants: Clinics
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Support | Medium Support | High Support | Comparison | Total
Number analyzed (Participants) | 3849 | 5098 | 3370 | 33638 | 45955
Number analyzed (Clinics) | 9 | 11 | 9 | 137 | 166
Age, Customized [Count of Participants; unit: Participants]
  18-21 years | 31 | 33 | 24 | 212 | 300
  22-39 years | 357 | 574 | 337 | 3649 | 4917
  40-75 years | 3169 | 4064 | 2744 | 27309 | 37286
  >75 years | 292 | 427 | 265 | 2468 | 3452
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2047 | 3057 | 1831 | 18707 | 25642
  Male | 1802 | 2041 | 1539 | 14931 | 20313
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Non-Hispanic white | 2417 | 880 | 2389 | 15582 | 21268
  Race/ethnicity: Non-Hispanic Black | 44 | 1364 | 196 | 7056 | 8660
  Race/ethnicity: Non-Hispanic Other | 127 | 350 | 126 | 2134 | 2737
  Race/ethnicity: Hispanic | 1249 | 2494 | 652 | 8734 | 13129
  Race/ethnicity: Unknown | 12 | 10 | 7 | 132 | 161

OUTCOME MEASURES:

1. Primary Outcome: Rate Ratio of the Percent of the Clinics' Patients "Indicated" for Statin With a Guideline-appropriate Prescription for Statins
Description: The data reported in the outcome measure data table is the rate ratio of the change in the percent of the clinic's 'indicated' patients with guideline-appropriate prescription for statins. Each monthly denominator included the patients who had an in-clinic encounter in the last year and were indicated for the medication per national guidelines that month. Therefore, the number of "participants" and who those "participants" were varied at each time of measurement. From month to month the set of "participants" could be completely different. The percent of patients indicated for a statin with an active prescription by month can be found in Figure 2 of the publication linked in this record: Gold, 2019. This is the only data available.
Time Frame: Monthly, up to 48 months
Population: The number of participants is not available for this study, only clinic-level data was collected.
Measure: Mean (95% Confidence Interval); unit: Rate ratio
Units Other Than Participants: Clinics
Arm/Group | Low Support | Medium Support | High Support | Comparison
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (Clinics) | 9 | 11 | 9 | 137
Rate ratio | 1.09 [1.06 to 1.13] | 1.11 [1.08 to 1.13] | 1.06 [1.03 to 1.09] | 1.04 [1.03 to 1.05]

2. Primary Outcome: Rate Ratio of the Percent of the Clinics' Patients "Indicated" for ACE/ARB With Guideline-appropriate Prescription for ACE/ARBs
Description: The data reported in the outcome measure data table is the rate ratio of the change in the percent of the clinic's 'indicated' patients with guideline-appropriate prescription for ACE/ARBs. Each monthly denominator included the patients who had an in-clinic encounter in the last year and were indicated for the medication per national guidelines that month. Therefore, the number of "participants" and who those "participants" were varied at each time of measurement. From month to month the set of "participants" could be completely different. The percent of patients indicated for an ACE/ARB with an active prescription by month can be found in Figure 3 of the publication linked in this record: Gold, 2019. This is the only data available.
Time Frame: Monthly, up to 48 months
Population: The number of participants is not available for this study, only clinic-level data was collected.
Measure: Mean (95% Confidence Interval); unit: Rate ratio
Units Other Than Participants: Clinics
Arm/Group | Low Support | Medium Support | High Support | Comparison
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (Clinics) | 9 | 11 | 9 | 137
Rate ratio | 0.95 [0.92 to 0.97] | 0.99 [0.97 to 1.01] | 0.99 [0.96 to 1.02] | 0.95 [0.94 to 0.95]

3. Secondary Outcome: Identify Clinic Characteristics Associated With the Support Strategies' Effectiveness (e.g. Decision-making Structures, Leadership Support, Team Processes I Characteristics, Readiness and Capacity for Change).
Description: Describe the characteristics of clinics that achieve sustained change and of those that do not achieve change
Time Frame: 3 years post-implementation
Reporting Status: Not Posted

4. Secondary Outcome: Rate Ratio of the Change in the Percent of the Clinic's 'Indicated' Patients With Correct Intensity Statin Prescribing
Description: The data reported in the outcome measure data table is the rate ratio of the change in the percent of the clinic's 'indicated' patients with correct intensity statin prescribing. Each monthly denominator included the patients who had an in-clinic encounter in the last year and were indicated for the medication per national guidelines that month. Therefore, the number of "participants" and who those "participants" were varied at each time of measurement. From month to month the set of "participants" could be completely different. The percent of patients with correct intensity statin prescribing by month can be found in Figure 2 of the publication linked in this record: Gold, 2019. This is the only data available.
Time Frame: Monthly, up to 48 months
Population: The number of participants is not available for this study, only clinic-level data was collected.
Measure: Mean (95% Confidence Interval); unit: Rate ratio
Units Other Than Participants: Clinics
Arm/Group | Low Support | Medium Support | High Support | Comparison
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (Clinics) | 9 | 11 | 9 | 137
Rate ratio | 1.24 [1.21 to 1.28] | 1.35 [1.31 to 1.39] | 1.11 [1.08 to 1.15] | 1.17 [1.16 to 1.18]

ADVERSE EVENTS:
Time Frame: No patients were recruited or consented in this study. Clinics were recruited and the intervention was conducted at the clinic level. With no patients enrolled we did not gather data on adverse events. Therefore there is not a time frame to report here.
Description: No patients were recruited or consented in this study. Clinics were recruited and the intervention was conducted at the clinic level. With no patients enrolled we did not gather data on adverse events.
Arm/Group | Low Support | Medium Support | High Support | Comparison
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT02325531/Prot_SAP_000.pdf